CLINICAL TRIAL: NCT03754829
Title: A Randomized Controlled Trial of a Web and Mobile Guided Psychological Intervention for Depressive Symptoms in Turkey.
Brief Title: Effectiveness of a Web and Mobile Guided Psychological Intervention for Depressive Symptoms in Turkey
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Burçin Ünlü İnce (Other)
Collaborators: Middle East Technical University (Other); VU University of Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Burçin Ünlü İnce, Ph.D., Postdoctoral Researcher, The Scientific and Technological Research Council of Turkey
Organization: The Scientific and Technological Research Council of Turkey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No: 53325897-115.02-E.263941
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Depressive Symptoms
Keywords: Randomized Controlled trial; Mobile Application; Problem-Solving Therapy; Online Guided Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A three-armed randomized controlled trial with 2 experimental groups and 1 control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSKA - Web Group (Experimental): The first experimental group will receive direct access to the web version of HSKA.
  Interventions: Behavioral: Her Sey Kontrol Altinda (HSKA)
- HSKA - Mobile Group (Experimental): The second experimental group will receive direct access to the mobile app of HSKA as well as automated supportive text messages based on PST.
  Interventions: Behavioral: Her Sey Kontrol Altinda (HSKA)
- Control Group (No Intervention): The control group consists of a wait-list and for ethical reasons, participants in this group will gain access to the intervention (either web or mobile application) four months after the baseline.

INTERVENTIONS:
Behavioral: Her Sey Kontrol Altinda (HSKA) — HSKA consists of 5 sessions over 5 weeks and is based on Problem-Solving therapy. Participants receive feedback on their homework assignments in brief weekly online messages from a clinical psychologist.
  Arms: HSKA - Mobile Group; HSKA - Web Group

SUMMARY:
The aim of this study is to test the clinical effects of a web and mobile application of guided Problem Solving Therapy for depressive symptoms among the general population in Turkey.

DETAILED DESCRIPTION:
In Turkey, there are serious deficiencies in mental health care. Among these, undertreatment of mentally ill patients, lack of psychologists and inadequate psychosocial and rehabilitation options for patients and their relatives are important prohibiting factors that reduce patients' outreach for getting help. While depression is highly prevalent (4.4%), only a small number of people seek professional help (18%) in Turkey. Innovative solutions are needed to overcome this treatment gap. Online Problem-Solving Therapy (PST) is a brief intervention proven to be effective in the treatment of depression, although little is known about its clinical effects in Turkey.

The aim of this study is to test the clinical effects of a web and mobile application of PST for depressive symptoms among the general population in Turkey.

Participants will be recruited through announcements in social media and the Middle East Technical University. A randomized controlled trial with a sample size of 444 participants randomized across three groups will be utilized. The first experimental group will receive direct access to the web version of the intervention; the second experimental group will receive direct access to the mobile app of the intervention as well as automated supportive text messages based on PST. The control group consists of a wait-list and for ethical reasons, participants in this group will gain access to the intervention (either web or mobile application) four months after the baseline. The intervention is based on an existing PST for the Turkish population, "Her Sey Kontrol Altinda" (HSKA).

ELIGIBILITY:
Inclusion Criteria:

* Turkish participants living in Turkey are eligible if the applicants are aged between 18-55 years and have mild to moderate depressive symptoms (Beck Depression Inventory-II score between 10 and 29).

Exclusion Criteria:

* Participants will be excluded if they have a BDI-II score above 29, or a medium-to- high suicidal risk (according to the MINI-International Neuropsychiatric Interview) and are advised to contact a psychiatrist or clinical psychologist.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 444 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Change on Beck Depression Inventory-II | Screening; baseline, 6-8 weeks after baseline and 4 months after baseline
  Depressive symptoms

SECONDARY OUTCOMES:
Change on State-Trait Anxiety Inventory (STAI) | baseline, 6-8 weeks after baseline and 4 months after baseline
  Anxiety symptoms
Change on Penn State Worry Questionnaire (PSWQ) | baseline, 6-8 weeks after baseline and 4 months after baseline
  The PSWQ will be used to measure pathological worry. It has 16 items in total. Each item can be scored on a five-point scale from 1 (not at all typical of me) to 5 (very typical of me), with a total score varying from 16 to 80. Higher scores indicating greater worry.
Change on Perceived Stress Scale (PSS) | baseline, 6-8 weeks after baseline and 4 months after baseline
  The PSS will be used to measure the perception of stress. It consists of 10 items for which the total score range is 0-40. Each item is rated on a five-point scale, from 0 (never) to 4 (very often). Higher scores indicating greater stress.
Change on General Self-Efficacy Scale (GSE) | baseline, 6-8 weeks after baseline and 4 months after baseline
  The GSE is a measure to assess self-efficacy beliefs. It contains 10 items, which are rated on a four-point scale from 1 (not at all true) to 5 (exactly true). The total score varies from 10 to 50. Higher scores indicating greater self-efficacy beliefs.
Change on EuroQol-5D-5L (EQ-5D-5L) | baseline, 6-8 weeks after baseline and 4 months after baseline
  EQ-5D-5L will be used to measure quality of life. It consists of 5 items each measuring different dimensions of health status (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The items are rated on a five-point scale from level 1 to level 5 (no problems; slight, moderate; severe and extreme problems). All the answers to each item are combined resulting in 3125 possible health states, ranging from 11111 (full health) to 55555 (worst health). Furthermore, there is a visual analogue scale (EQ-VAS) measuring a global rating of self-perceived health. This is scored by 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Satisfaction with the intervention questionnaire | 6-8 weeks after baseline only in the two experimental groups
  Participants will be asked about each module to define their satisfaction with the module concerned ('Was this lesson useful to you?'). The answers can be rated on a 5-point Likert scale from 1 (not at all) to 5 (very useful).

OTHER OUTCOMES:
MINI-International Neuropsychiatric Interview | Screening
  Suicidal ideations

CONTACTS AND LOCATIONS:
Locations (1):
- Middle East Technical University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Unlu Ince B, Gokcay D, Riper H, Cuijpers P. Effectiveness of a Web- and Mobile-Guided Psychological Intervention for Depressive Symptoms in Turkey: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Apr 5;8(4):e13239. doi: 10.2196/13239. PMID 30950802